CLINICAL TRIAL: NCT05248646
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Sibeprenlimab Administered Subcutaneously in Subjects With Immunoglobulin A Nephropathy.
Brief Title: Visionary Study: Phase 3 Trial of Sibeprenlimab in Immunoglobulin A Nephropathy (IgAN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 417-201-00007
Record Dates: First submitted 2022-02-18; First posted 2022-02-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: IgAN; Sibeprenlimab; VIS649
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sibeprenlimab 400 mg s.c. q 4weeks (Active Comparator)
  Interventions: Drug: Sibeprenlimab 400 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sibeprenlimab 400 mg — Sibeprenlimab 400 mg s.c. q 4 weeks
  Other Names: VIS649
  Arms: Sibeprenlimab 400 mg s.c. q 4weeks
Drug: Placebo — Placebo s.c. q 4 weeks
  Arms: Placebo

SUMMARY:
This is a phase 3 study to evaluate effects on proteinuria and glomerular filtration rate of sibeprenlimab 400 mg subcutaneously (s.c.) Q 4 weeks in adults with IgAN who are receiving maximally tolerated standard-of-care therapy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of sibeprenlimab 400 mg administered SC Q 4 weeks compared to placebo in patients with IgAN. The primary objective is to compare the relative change from baseline in the urinary protein to creatinine ratio (uPCR) in 24-hour urine collections, after 9 months of treatment. The key secondary objective is to compare the annualized rate of change from baseline (slope) of estimated glomerular filtration rate (eGFR) after approximately 24 months of treatment. There will be one main cohort comprised of approximately 450 subjects with source-verified biopsy-confirmed IgAN and eGFR ≥ 30 mL/min/1.73 m^2. An additional exploratory cohort will be comprised of up to 20 subjects with source-verified biopsy confirmed IgAN and eGFR of 20 to < 30 mL/min/1.73 m^2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age .
* Biopsy-confirmed IgAN. (Patients with an eGFR of 30 to 45 mL/min/1.73m2 must have had a kidney biopsy performed within 36 months of the screening visit).
* Stable and maximally tolerated dose of ACEI and/or ARB for at least 3 months prior to screening. Patients who are on a stable dose of SGLT2i may participate if treatment was initiated ≥3 months prior to screening. Patients who are unable to take an ACEI or ARB may participate if their overall management conforms with standards of care and other protocol requirements.
* Screening urine protein/creatinine ratio (uPCR) ≥ 0.75 g/g or urine protein ≥ 1.0 g/day
* eGFR ≥ 30 mL/min/1.73 m2, (for the exploratory cohort only: eGFR 20- <30 mL/min/1.73 m2), calculated using the CKD-EPI equation.)

Exclusion Criteria:

* Secondary forms of IgAN or IgA vasculitis.
* Coexisting chronic kidney disease other than IgAN.
* Kidney biopsy findings in addition to IgAN including those of diabetic nephropathy, membranous nephropathy, or lupus nephritis. Hypertensive vascular changes are acceptable.
* Kidney biopsy MEST or MEST-C score of T2 or C2 (Oxford IgAN classification). If MEST-scoring was not performed, the presence of > 50% tubulo-interstitial fibrosis, or crescents in > 25% of glomeruli is exclusionary. This does not apply to the exploratory cohort.
* Nephrotic syndrome
* Serum IgG < 600 mg/dL at screening.
* Chronic systemic immunosuppression, including glucocorticoids, within 16 weeks of randomization
* Participation in another interventional clinical trial and receipt of another investigational drug within 30 days prior to the administration of IMP or 5 half-lives from last investigational drug administration, whichever is longer.
* Chronic infectious disease, or acute infectious disease at time of screening.
* Type 1 diabetes, or poorly controlled Type 2 diabetes
* Uncontrolled hypertension

The protocol provides additional information about these and other inclusion and exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Urinary protein to creatinine ratio (uPCR) in a 24-hour collection | At 9 months

SECONDARY OUTCOMES:
Annualized rate of change from baseline (slope) of eGFR | Over 24 months
Proportion of subjects achieving urine total protein < 1.0 g/day and ≥ 25% reduction from baseline. | At 12 months
Annualized slope of eGFR | Over 12 months

CONTACTS AND LOCATIONS:
Locations (297):
- United States (48):
  - University of Alabama at Birmingham - Site #336, Birmingham, Alabama
  - Mayo Clinic Arizona - Site #363, Phoenix, Arizona
  - University of Arkansas for Medical Sciences - Site #353, Little Rock, Arkansas
  - Amicis Research Center - Site #341, Granada Hills, California
  - University of CA San Diego - Site #351, La Jolla, California
  - California Institute of Renal Research - Site #371, La Mesa, California
  - Loma Linda University Health Care Clinical Trial Center Clinic - Site #372, Loma Linda, California
  - Academic Medical Research Institute - Site #333, Los Angeles, California
  - Kaiser Permanente - Southern California Permanente Medical Group SCPMG - LAMC - Site #325, Los Angeles, California
  - Stanford University - Site #370, Palo Alto, California
  - North America Research Institute - Site #335, San Dimas, California
  - University of California, San Francisco - Site #377, San Francisco, California
  - Colorado Kidney Care PC - Site #330, Denver, Colorado
  - Mayo Clinic in Florida - Site #321, Jacksonville, Florida
  - South Florida Research Institute - Site #323, Lauderdale Lakes, Florida
  - Columbus Research Group - Site #376, South Miami, Florida
  - Fides Clinical Research North Atlanta Kidney Specialists - Site #373, Atlanta, Georgia
  - Georgia Nephrology - Site #356, Lawrenceville, Georgia
  - University of Iowa Hospitals & Clinics - Site #359, Iowa City, Iowa
  - Kansas Nephrology Associates - Site #322, Wichita, Kansas
  - Ochsner Medical Center - Site #334, New Orleans, Louisiana
  - University of Maryland - Site #355, Baltimore, Maryland
  - MGH Harvard - Site #369, Boston, Massachusetts
  - Brigham and Women's Hospital, Division of Renal Medicine - Site #379, Boston, Massachusetts
  - Tufts Medical Center - Site #349, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Site #337, Boston, Massachusetts
  - UMASS Memorial Medical Center - Site #331, Worcester, Massachusetts
  - St. Clair Nephrology Research - Site #320, Roseville, Michigan
  - University of Minnesota - Site #345, Minneapolis, Minnesota
  - Mayo Clinic - Rochester - Site #332, Rochester, Minnesota
  - University of Nebraska Medical Center - Site #347, Omaha, Nebraska
  - Davita Clinical Research - Las Vegas - Site #327, Las Vegas, Nevada
  - Northwell Health - North Shore University Hospital NSUH - Site #346, Great Neck, New York
  - New York University Grossman School of Medicine - Site #362, New York, New York
  - Jacobi Medical Center - Site #364, The Bronx, New York
  - The University of Cincinnati - Site #343, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center - Site #350, Columbus, Ohio
  - Rhode Island Hospital - Site #367, Providence, Rhode Island
  - Dunes Clinical Research LLC - Site #374, Dakota Dunes, South Dakota
  - Research Management, Inc - Site #354, Austin, Texas
  - Renal Disease Research Institute - Site #378, Dallas, Texas
  - Baylor College of Medicine (BCM) Medical Center - Site #375, Houston, Texas
  - Prolato Clinical Research Center (PCRC) - Site #324, Houston, Texas
  - Pioneer Research Solutions, Inc. - Site #339, Houston, Texas
  - UT Health Science Center at San Antonio - Site #368, San Antonio, Texas
  - Utah Kidney Research Institute - Site #342, Salt Lake City, Utah
  - University of Wisconsin - Site #352, Madison, Wisconsin
  - Medical College of Wisconsin - Site #361, Milwaukee, Wisconsin
- Argentina (4):
  - Hospital Britanico de Buenos Aires - Site #800, Buenos Aires
  - Maffei Centro Medico - Site #802, Buenos Aires
  - Clinica Privada Velez Sarsfield - Nephrology and Transplantation Service - Site #801, Córdoba
  - Centro de Salud Renal Junin S.R.L. - Site #803, Junín
- Australia (14):
  - Canberra Hospital - Site #3, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital (CRGH) (Concord Hospital) - Site #13, Concord, New South Wales
  - St. George Hospital - Site #14, Kogarah, New South Wales
  - University of New South Wales (UNSW) - Liverpool Hosp - Site #11, Liverpool, New South Wales
  - John Hunter Hospital - Site #5, New Lambton Heights, New South Wales
  - Prince of Wales Hospital - Site #2, Randwick, New South Wales
  - Royal North Shore Hospital - Site #6, Saint Leonards, New South Wales
  - Royal Adelaide Hospital - Site #12, Adelaide, South Australia
  - Flinders Medical Centre - Site #9, Bedford Park, South Australia
  - Launceston General Hospital - Site #8, Launceston, Tasmania
  - The University of Melbourne - St. Vincent's Hospital Melbourne (SVHM) - Site #1, Fitzroy, Victoria
  - Western Health Sunshine Hospital - Site #10, St Albans, Victoria
  - Fiona Stanley Hospital (FSH) - Site #4, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital - Site #7, Nedlands, Western Australia
- Belgium (5):
  - Hopital Erasme - Site #402, Brussels
  - UZ Leuven Campus Gasthuisberg - Site #401, Genk
  - Ziekenhuis Oost Limburg Genk ZOL - Site #405, Genk
  - AZ Sint Lucas - Site #403, Ghent
  - CHR de la Citadelle - Site #400, Liège
- Brazil (11):
  - Universidade Federal do CearClinic Pro-nefron - Site #827, Fortaleza, Ceará
  - Clinica Senhor do Bonfim Ltda CSB - Monte Serrat - Site #826, Salvador, Estado de Bahia
  - Recife - Site #820, Recife, Pernambuco
  - Santa Casa de Misericordia - Porto Alegre - Site #824, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre HCPA - Site #828, Porto Alegre, Rio Grande do Sul
  - Fundacao Pro Rim - Site #821, Joinville, Santa Catarina
  - Centro de Pesquisa Medica Praxis - Site #825, Santo André, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto - SP FAMERP - Hospital de Base HB - Site #822, São José do Rio Preto, São Paulo
  - Universidade de Sao Paulo (USP) - Faculdade de Medicina (FMUSP) - Site #823, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - Escola Paulista de Medicina EPM - Hospital do Rim e Hipertensao HRIM - Site #830, São Paulo, São Paulo
  - Universidade estadual do Rio de Janeiro - Site #831, Rio de Janeiro
- Canada (8):
  - University of Calgary - Health Research Innovation Centre: Sheldon Chumir Health Centre - Site #300, Calgary, Alberta
  - St. Joseph's Healthcare Hamilton - Site #307, Hamilton, Ontario
  - Clinical Research Solutions Inc. - Site #301, Kitchener, Ontario
  - Lakeridge Health Oshawa - Site #303, Oshawa, Ontario
  - OTT Healthcare Inc. - Site #305, Scarborough Village, Ontario
  - Office of Stephen S. Chow, MD - Site #306, Toronto, Ontario
  - CISSS de la Monteregie centre-Centre de recherche Hopital Charles Lemoyne - Site #302, Greenfield Park, Quebec
  - McGill University Health Centre - Site #304, Montreal, Quebec
- China (25):
  - Capital Medical University (CMU) - Beijing Anzhen Hospital (BAH) - Site #36, Beijing, Beijing Municipality
  - Peking University People's Hospital - Site #32, Beijing, Beijing Municipality
  - Peking University First Hospital - Site #20, Beijing, Beijing Municipality
  - Peking University International Hospital - Site #34, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital - Site #33, Beijing, Beijing Municipality
  - Xiamen University - Zhongshan Hospital - Site #42, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital - Site #39, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat - sen University - Site #40, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University - Site #28, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital - Site #43, Shenzhen, Guangdong
  - Liuzhou Workers Hospital - Site #35, Liuchow, Guangxi
  - The Peoples Hospital of Guangxi zhuang Autonomous Region - Site #27, Nanning, Guangxi
  - Renmin Hospital of Wuhan University - Site #24, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University - Site #44, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical University - Site #29, Baotou, Inner Mongolia Proviance
  - Wuxi Peoples' Hospital affiliated to Nanjing Medical University - Site #30, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University - Site #22, Nanchang, Jiangxi
  - Jiangxi Pingxiang Peoples' Hospital - Site #21, Pingxiang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University - Site #31, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical College - Site #23, Xi'an, Shaanxi
  - The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) - Site #26, Jinan, Shandong
  - Yantai Yuhuangding Hospital - Site #41, Yantai, Shandong
  - Sichuan Provincial Peoples Hospital - Site #38, Chengdu, Sichuan
  - Yibin Second Peoples Hospital - Site #25, Yibin, Sichuan
  - Zhejiang Provincial People's Hospital - Site #37, Hangzhou, Zhejiang
- Croatia (4):
  - University Hospital Center Osijek - Site #410, Osijek
  - University Hospital Center Split - Site #413, Split
  - Klinicka Bolnica Dubrava (KBD) (Clinical Hospital Dubrava) - Site #411, Zagreb
  - University Hospital Merkur - Site #414, Zagreb
- Vseobecna fakultni nemocnice v Praze - Site #420, Prague, Czechia
- France (14):
  - Hopital Pellegrin - Site #431, Bordeaux, Aquitaine
  - CHU de Grenoble Alpes - Hopital Nord Michallon - Site #433, Grenoble, Auvergne-Rhône-Alpes
  - CHU Clermont-Ferrant-Gabriel Montpied - Site #443, Clermont-Ferrand, Auvergne
  - CHU de Reims Hopital Maison Blanche - Site #442, Reims, Champagne-Ardenne
  - Centre Hospitalier Universitaire de Nimes CHU - Hopital Universitaire Caremeau - Site #430, Nîmes, Gard
  - Hopital Emile Muller - Site #438, Mulhouse, Haut-Rhin
  - CHU Amiens-Picardie Nephrology Dialysis Transplantation - Site #440, Amiens, Hauts-de-France
  - CHU Hotel Dieu, Nephrologie - Immunologie clinique - Transplantation - Site #432, Nantes, Loire-Atlantique
  - CH Limoges - Site #439, Limoges, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Saint-Etienne - Hopital Nord - Site #434, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier Henri Duffaut - Site #441, Avignon, Provence-Alpes-Côte d'Azur Region
  - Hopital La Conception Centre de Nephrologie et de Transplantation Renal - Site #437, Marseille, Provence-Alpes-Côte d'Azur Region
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopitaux Universitaires Henri Mondor (Hopital Henri-Mondor) - Site #436, Créteil, Île-de-France Region
  - Hopital de Tenon Sorbonne Universite - Site #435, Paris, Île-de-France Region
- Germany (4):
  - Agaplesion Markus Krankenhaus - Site #457, Frankfurt am Main, Hesse
  - DaVita Clinical Research Germany GmbH - Site #456, Düsseldorf, North Rhine-Westphalia
  - Universitaetsmedizin Mainz - Site #455, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus - Site #450, Dresden, Saxony
- Greece (6):
  - Hippokration General Hospital of Athens, Nephrology Clinic - Site #475, Athens
  - Nephrology Department, University General Hospital of Heraklion - Site #472, Heraklion
  - University Hospital of Ioannina (UHI) - Nephrology Clinic - Site #471, Ioannina
  - University of Thessaly, Nephrology Clinic - Site #474, Larissa
  - Aristotle University of Thessaloniki (AUTH) - Hippokration Hospital - Site #470, Thessaloniki
  - Hellenic Republic Ministry of Health & Welfare - General Hospital of Thessaloniki (George Papanikolaou) - Site #473, Thessaloniki
- Hong Kong (5):
  - Queen Mary Hospital - Site #60, Hong Kong
  - Tung Wah Hospital - Site #61, Hong Kong
  - Princess Margaret Hospital - Site #62, Kowloon
  - Prince of Wales Hospital - Site #63, Shatin
  - Yan Chai Hospital - Site #64, Tsuen Wan
- Hungary (2):
  - Pecsi Tudomanyegyetem, Altalanos Orvostudomanyi KarKlinikai Kozpont II - Site #482, Pécs, Baranya
  - Somogy Megyei Kaposi Mor Oktatokorhaz - Site #481, Kaposvár, Somogy County
- India (15):
  - Kusum Dhirajlal Hospital - Site #73, Ahmedabad, Gujarat
  - Muljibhai Patel Urological Hospital (MPUH) (Kidney Hospital) - Site #70, Nadiād, Gujarat
  - M.S. Ramaiah Memorial Hospital - Site #72, Bengaluru, Karnataka
  - Mazumdar Shaw Medical Centre - A unit of Narayana Health - Site #87, Bengaluru, Karnataka
  - Manipal University - Kasturba Medical College - Site #79, Manipal, Karnataka
  - Government Medical College - Site #71, Kozhikode, Kerala
  - Government Medical College Thiruvananthapuram - Site #74, Thiruvananthapuram, Kerala
  - Mahatma Gandhi Mission Institute of Health Scienes MGMIHS - Mahatma Gandhi Mission MGM Medical Centre Research Institute - Aurangabad - Site #82, Aurangabad, Maharashtra
  - Life Point Multispecialty Hospital - Site #84, Pune, Maharashtra
  - Sir Ganga Ram Hospital - Site #75, New Delhi, National Capital Territory of Delhi
  - Postgraduate Institute of Medical Education Research PGIMER - Site #77, Chandigarh, Punjab
  - Christian Medical College & Hospital (CMCH) - Vellore - Site #80, Vellore, Tamil Nadu
  - Osmania General Hospital (OGH) - Site #78, Hyderabad, Telangana
  - Nizams Institute of Medical Sciences NIMS - Site #81, Hyderabad, Telangana
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS) - Site #76, Lucknow, Uttar Pradesh
- Israel (6):
  - The Barzilai Medical Center (The Ashkelon Hospital) - Site #494, Ashkelon
  - Technion-Israel Institute of Technology - The Lady Davis Carmel Medical Center (LDCMC) - Institute of Nephrology and Hypertension - Site #491, Haifa
  - Shaare Zedek Medical Center (SZMC) - Site #492, Jerusalem
  - Tel Aviv University Sackler School of Medicine - Meir Medical Center (MMC) (Meir Hospital) - Site #490, Kfar Saba
  - Galilee Medical Center (Western Galilee Hospital) - Site #495, Nahariya
  - Rabin Medical Center - Institute of Nephrology and Hypertension - Diabetic Nephropathy Clinic - Site #493, Petah Tikva
- Italy (13):
  - IRCCS Azienda Ospedaliero-Universitaria Policlinico Sant Orsola - Site #512, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia - Site #504, Brescia
  - Azienda Ospedaliero-Universitaria Careggi Firenze - Site #500, Florence
  - Ospedale San Giovanni di Dio - Site #506, Florence
  - Clinica Nefrologica, Dialisi e Trapianto, IRCCS Ospedale Policlinico San Martino - Site #503, Genova
  - AOU Gaetano Martino di Messina U.O.C., Nefrologia e Dialisi - Site #502, Messina
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico - Site #513, Milan
  - Campania Luigi Vanvitelli - Site #510, Napoli
  - Fondazione Maugeri - Site #509, Pavia
  - AUSL Hospital Guglielmo da Saliceto - Site #507, Piacenza
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Site #501, Roma
  - ULSS 6 Vicenza - Ospedale San Bortolo di Vicenza - Site #505, Vicenza
  - Ospedale di Belcolle Viterbo - Site #514, Viterbo
- Japan (30):
  - Nagoya University Hospital - Site #705, Nagoya, Aichi-ken
  - Fujita Health University Hospital - Site #709, Toyoake, Aichi-ken
  - Juntendo University - Urayasu Hospital - Site #707, Urayasu, Chiba
  - Kurume University Hospital - Site #725, Kurume, Fukuoka
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC) - Site #723, Amagasaki, Hyōgo
  - Kobe University Hospital - Site #724, Kobe, Hyōgo
  - University of Tsukuba Hospital - Site #708, Tsukuba, Ibaraki
  - Kanazawa University Hospital - Site #702, Kanazawa, Ishikawa-ken
  - Toranomon Hospital Kajigaya - Site #714, Kawasaki, Kanagawa
  - Kitasato University Hospital - Site #729, Sagamihara, Kanagawa
  - Tohoku Medical and Pharmaceutical University Hospital - Site #718, Sendai, Miyagi
  - Nara Medical University Hospital - Site #713, Kashihara, Nara
  - Juntendo University Nerima Hospital - Site #727, Tokyo, Nerima-ku
  - Oita University Hospital - Site #717, Yufu, Oita Prefecture
  - Osaka University Hospital - Site #719, Suita, Osaka
  - Hamamatsu University Hospital - Site #704, Hamamatsu, Shizuoka
  - Japanese Red Cross Ashikaga Hospital - Site #726, Ashikaga, Tochigi
  - Juntendo University Hospital - Site #715, Bunkyō-Ku, Tokyo
  - The Jikei University Hospital - Site #712, Minato-Ku, Tokyo
  - Tokyo Medical University Hospital - Site #728, Shinjuku-Ku, Tokyo
  - Tokyo Women's Medical University Hospital - Site #710, Shinjuku-Ku, Tokyo
  - Teikyo University Hospital - Site #706, tabashi City, Tokyo
  - NHO Chibahigashi National Hospital - Site #700, Chiba
  - Kyushu University Hospital (KUH) - Site #703, Fukuoka
  - Fukuoka University - Fukuoka University Hospital - Site #722, Fukuoka
  - University of Miyazaki Hospital - Site #716, Miyazaki
  - Nagasaki University Hospital - Site #720, Nagasaki
  - Niigata University Medical & Dental Hospital - Site #711, Niigata
  - Okayama University Hospital - Site #701, Okayama
  - Osaka General Medical Center - Site #721, Osaka
- Malaysia (7):
  - Hospital Kuala Lumpur - Site #123, Kuala Lumpur, Kuala Lumpur
  - Hospital Canselor Tuanku Muhriz UKM - Site #125, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre - Site #121, Kuala Lumpur, Kuala Lumpur
  - Hospital Tuanku Ja'afar - Site #122, Seremban, Negeri Sembilan
  - Hospital Tengku Ampuan Afzan - Site #120, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun - Site #124, Ipoh, Perak
  - Sunway Medical Centre (SMC) - Site #126, Petaling Jaya, Selangor
- Netherlands (4):
  - Radboud Universitair Medisch Centrum - Site #520, Nijmegen, Gelderland
  - Maastricht University Medical Center (MUMC) - Site #523, Maastricht, Limburg
  - Groene Hart Ziekenhuis, Ioc, Bleuland - Site #521, Gouda, South Holland
  - Amsterdam UMC - Site #522, Amsterdam
- Philippines (3):
  - University of Santo Tomas Hospital - Site #130, Manila
  - National Kidney Institute - Site #132, Quezon
  - St. Luke's Medical Center - Quezon City - Site #131, Quezon
- Poland (4):
  - Uniw. Szp. Kliniczny w Bialymstoku, 2nd Department of Nephrology and Hypertension with Dialysis Unit - Site #531, Bialystok, Bialystok
  - Szpital Uniwersytecki w Krakowie - Site #533, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne PROMED - Site #535, Krakow, Malopotskie
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w odzi - Site #530, Lodz, Łódź Voivodeship
- Portugal (5):
  - Centro Clinico Academico - Braga - Site #540, Braga
  - Centro Hospitalar de Lisboa Ocidental (CHLO), E.P.E. - Hospital de Santa Cruz (HSC) - Site #545, Carnaxide
  - Hospital Beatriz Angelo (HBA) - Site #541, Lisbon
  - Servico de Nefrologia - Centro Hospitalar Universitario Sao Joao (CHUSJ), EPE - Site #544, Porto
  - Centro Hospitalar de Vila Nova de Gaia / Espinho - Site #543, Porto
- Singapore (3):
  - National University Hospital - Site #142, Singapore, Central Singapore
  - Singapore General Hospital (SGH) - Site #141, Singapore, Central Singapore
  - Tan Tock Seng Hospital - Site #140, Singapore, Central Singapore
- South Korea (14):
  - Pusan National University Hospital - Site #102, Busan, Busan Gwang'yeogsi
  - Kyungpook National UniversityA Hospital - Site #112, Daegu, Daegu Gwang'yeogsi
  - Chonnam National University Hospital - Site #113, Gwangju, Gwangiu Gwang'yeogsi
  - National Health Insurance Service Ilsan Hospital - Site #114, Goyang-si, Gyeonggi-do
  - Hallym University Medical Center - Sacred Heart Hospital - Site #104, Anyang, Gyeonggido
  - Hallym University Medical Center - Dongtan Sacred Heart Hospital - Site #109, Hwasŏng, Gyeonggido
  - Seoul National University Bundang Hospital - Site #110, Seongnam, Gyeonggido
  - Asan Medical Center (AMC) - Site #111, Seoul, Seoul Teugbyeoisi
  - Kyung Hee University International Medical Service Gangdong Kyung Hee University KHU - Site #105, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital - Site #107, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center - Site #108, Seoul, Seoul Teugbyeolsi
  - Kangdong Sacred Heart Hospital - Site #106, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Site #100, Seoul, Seoul Teugbyeolsi
  - Yonsei University Severance Hospital - Site #103, Seoul, Seoul Tukpyolshi
- Spain (14):
  - Hospital Universitario de A Corua - Site #569, A Coruña
  - Hospital Universitario Cruces - Site #574, Barakaldo
  - Hospital del Mar - Site #572, Barcelona
  - Fundacio Puigvert - Site #567, Barcelona
  - Hospital Universitari Vall d'Hebron - Site #566, Barcelona
  - Hospital Universitari de Bellvitge - Site #563, Barcelona
  - Hospital Clinico San Carlos - Site #564, Bilbao
  - Hospital Universitario Reina Sofia - Site #565, Córdoba
  - Hospital Arquitecto Marcide de Ferrol - Site #575, Ferrol
  - Hospital Universitario Puerta de Hierro - Site #570, Madrid
  - Hospital Universitario Marques de Valdecilla - Site #560, Santander
  - Hospital Universitario Virgen Macarena - Site #562, Seville
  - Hospital Universitario Virgen del Rocio - Site #561, Seville
  - Hospital Universitario Dr. Peset - Site #568, Valencia
- Sri Lanka (5):
  - National Hospital of Sri Lanka - Site #151, Colombo
  - Karapitiya Teaching Hospital - Site #153, Galle
  - National Hospital Kandy - Site #152, Kandy
  - Kurunegala Teaching Hospital - Site #154, Kurunegala
  - Sri Jayewardenepura General Hospital (SJGH) - Site #150, Nugegoda
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital - Site #161, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital - Site #160, Keelung
  - Shuang Ho Hospital - Site #163, New Taipei City
  - Taichung Veterans General Hospital - Site #162, Taichung
  - National Taiwan University Hospital - Site #164, Taipei
  - Taipei Veterans General Hospital - Site #165, Taipei
- Thailand (6):
  - Navamindradhiraj University - Site #174, Bangkok
  - King Chula Memorial Hospital, Chulalongkorn University - Site #170, Bangkok
  - Phramongkutklao Hospital - Site #175, Bangkok
  - Ramathibodi Hospital - Site #171, Bangkok
  - Chiang Mai University - Site #172, Chiang Mai
  - Khon Kaen University - Site #173, Khon Kaen
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust - Site #580, Cambridge
  - Gloucestershire Royal Hospital - Site #586, Gloucester
  - University Hospitals of Leicester NHS Trust - Site #581, Leicester
  - Barts Health NHS Trust - The Royal London Hospital - Site #584, London
  - Royal Free Hospital London NHS Trust - Site #585, London
  - King's College Hospital, NHS Foundation Trust - Site #582, London
  - Salford Royal NHS Foundation Trust - Site #583, Salford
  - Clinical Research Unit, Morriston Hospital - Site #588, Swansea
- Vietnam (3):
  - Viet Duc Hospital - Site #181, Hanoi
  - Nguyen Tri Phuong Hospital - Site #180, Ho Chi Minh City
  - Hue Central Hospital - Site #182, Huế

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Perkovic V, Barratt J, Lafayette R, Liew A, Suzuki Y, Carroll K, Cheung CK, Tesar V, Trimarchi H, Wong MG, Zhang H, Xia J, Fajardo C, Shah L, Hafkin J, Rizk DV. Evaluating Sibeprenlimab in IgA Nephropathy - Rationale and Baseline Data from the VISIONARY Trial. Kidney Int Rep. 2025 Oct 1;10(12):4207-4218. doi: 10.1016/j.ekir.2025.09.031. eCollection 2025 Dec. PMID 41426046
- [Derived] Perkovic V, Trimarchi H, Tesar V, Lafayette R, Wong MG, Barratt J, Suzuki Y, Liew A, Zhang H, Carroll K, Jha V, Quevedo A, Han SH, Praga M, Chacko B, Sahay M, Cheung CK, Kooienga L, Walsh M, Xia J, Fajardo C, Shah L, Hafkin J, Rizk DV; VISIONARY Trial Investigators Group. Sibeprenlimab in IgA Nephropathy - Interim Analysis of a Phase 3 Trial. N Engl J Med. 2025 Nov 8. doi: 10.1056/NEJMoa2512133. Online ahead of print. PMID 41211929
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397